CLINICAL TRIAL: NCT05003505
Title: Characteristics of Vaginal and Intestinal Microbiota in Women With Different Cervical HPV Infection
Brief Title: Characteristics of Vaginal and Intestinal Microbiota and Cervical HPV Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Binhua Dong, Laboratory of Gynecologic Oncology, Fujian Maternity and Child Health Hospital
Other Study IDs: CVMC2018
Record Dates: First submitted 2021-07-12; First posted 2021-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intestinal Microbiota; Vaginal Microbiota; HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — DNA specimens of exfoliated cervix cells；DNA samples of vaginal secretions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with cervical cytology (TCT) abnormalities: In the enrollment, women who have undergone cervical cytology (TCT) examination for the last 3 months with abnormal results will be included in this study. All participants will be followed up three times, at 6 months, 12 months and 24 months.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Participants will be followed up at 6, 12 and 24 months with the test of enous blood, vaginal secretions, faeces, and cervical exfoliated cells.

SUMMARY:
There are different microbial communities on the surface of human body (skin, hair, nails, etc.) and in the cavity connected with the outside world. The human microbiota is the general term of the genetic information of microorganisms that coexist with human beings and cause various diseases under certain conditions. The results of human microbial genome analysis show that the microbial communities in different parts of the human body and different individuals have amazing diversity, some of which play an important role in human health, and some are closely related to diseases. Female lower genital tract infection is often associated with human papillomavirus (HPV) infection and bacterial vaginosis (BV), such as cervical and vaginal precancerous lesions, cancer, condyloma acuminatum and other sexually transmitted diseases (STD). Persistent infection of high-risk human papillomavirus (HR-HPV) is closely related to the occurrence of invasive cervical cancer. New evidence suggests that vaginal microbiota composition is different in women with HR-HPV infection and high-grade cervical lesions. The increase of the severity of cervical intraepithelial neoplasia is related to the decrease of the relative abundance of vaginal Lactobacillus. In addition to vaginal microbes, the powerful intestinal flora is considered to be the "invisible organ" of the human body. There is a dynamic and balanced interaction network between intestinal microorganisms and human immune cells. Once the intestinal flora is out of balance, the changes in species, quantity, proportion, location and biological characteristics will cause a series of inflammatory reactions and immune system diseases, and even lead to cancer. Some studies have shown that there is a potential relationship between intestinal microorganisms and vaginal microorganisms. Recent research evidence suggests that the mutually beneficial relationship between oral bacteria and other vaginal bacteria supports the colonization of pathogens and may help maintain the characteristics of vaginal flora imbalance.

DETAILED DESCRIPTION:
Based on the clinical practice, this study carried out a multi center cohort study in Fujian Province, China. In this study, five research including Fujian Maternity and Child Health Hospital, Mindong Hospital of Ningde City, Zhangzhou affiliated Hospital of Fujian Medical University, Quanzhou First Hospital Afflicated to Fujian Medical University and Xiamen Maternity and Child Health Hospital Affiliated to Xiamen University were included, each of which included 600 individuals, with a total of 3000 women with potential cervical lesions were enrolled. Blood samples were tested for immunology, stool swabs and vaginal secretions were collected for microecological evaluation. At the same time, 21 kinds of common HPV virus types, cervical exfoliative cytology and 10 kinds of common STDs pathogens were detected. The included population will be tested with the same samples at 6, 12 and 24 months of follow-up to explore the relationship between vaginal, intestinal microorganisms and cervical HPV infection and the development of cervical lesions and its potential impact, so as to further explore the key factors affecting the persistent infection and clearance of HPV in female reproductive tract and the potential impact factors of the occurrence and development of cervical lesions. This prospective observational the characteristics of vaginal and intestinal microbiota in women with different cervical HPV infection, to evaluate the relationship and the underlying effect in the developoing of cervical lessions.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-65.
* TCT examination was performed in the last 3 months with abnormal results.
* Non pregnant people with sexual history.
* Asexual life, no vaginal medication or flushing before 72 hours of sampling.

Exclusion Criteria:

* Within 8 weeks after pregnancy or postpartum.
* Patients with history of genital tract tumor.
* History of HPV vaccination.
* Previous history of hysterectomy, cervical surgery, pelvic radiotherapy Historical.
* In recent one month, she has received genital tract infection, HPV or other STDs treatment related to the infection of mycoplasma.
* Use antibiotics or vaginal microecological improvement products in recent 1 month.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese women aged 20-65 years with abnormal cervical cytology.
Sampling Method: Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical histopathology testing at baseline | Baseline
  Cervical histopathology was performed at baseline for all participants.
Cervical histopathology testing at 12-month follow-up | 12-month follow-up
  Cervical histopathology was performed at 12-month follow-up for cervical HPV infection or cytology abnormalities women.
Cervical histopathology testing at 24-month follow-up | 24-month follow-up
  Cervical histopathology was performed at 24-month follow-up for cervical HPV infection or cytology abnormalities women.
Human Papillomavirus (HPV) DNA testing at baseline | baseline
  All participants were tested for HPV DNA of cervical exfoliated cells at the time of baseline.
Human Papillomavirus (HPV) DNA testing at 6-month follow-up | 6-month follow-up
  All participants were tested for HPV DNA of cervical exfoliated cells at the time of 6-month follow-up.
Human Papillomavirus (HPV) DNA testing at 12-month follow-up | 12-month follow-up
  All participants were tested for HPV DNA of cervical exfoliated cells at the time of 12-month follow-up.
Human Papillomavirus (HPV) DNA testing at 24-month follow-up | 24-month follow-up
  All participants were tested for HPV DNA of cervical exfoliated cells at the time of 24-month follow-up.
Cervical cytology testing at baseline | baseline
  All participants were tested for cervical cytology at the time of baseline.
Sequencing of the vaginal microbiota at baseline | baseline
  All participants underwent microbiological metagenomic sequencing of vaginal secretions at baseline.
Sequencing of the vaginal microbiota at 6-month follow-up | 6-month follow-up
  All participants underwent microbiological metagenomic sequencing of vaginal secretions at 6-month follow-up.
Sequencing of the vaginal microbiota at 12-month follow-up | 12-month follow-up
  All participants underwent microbiological metagenomic sequencing of vaginal secretions at 12-month follow-up.
Sequencing of the vaginal microbiota at 24-month follow-up | 24-month follow-up
  All participants underwent microbiological metagenomic sequencing of vaginal secretions at 24-month follow-up.
Sequencing of the gut microbiota at baseline | baseline
  All participants underwent fecal microbiome sequencing at baseline.
Sequencing of the gut microbiota at 6-month follow-up | 6-month follow-up
  All participants underwent fecal microbiome sequencing at 6-month follow-up.
Sequencing of the gut microbiota at 12-month follow-up | 12-month follow-up
  All participants underwent fecal microbiome sequencing at 12-month follow-up.
Untargeted Metabolites of vaginal secretions testing at baseline | baseline
  All participants were tested for microbial untargeted metabolites of vaginal secretions at baseline by liquid chromatography tandem mass spectrometric (LC-MS). Measure abundances of vaginal secretions metabolites, metabolic networks, and metabolic pathways activity.
Change in vaginal secretions metabolome from baseline to 12-month follow-up assessments | 6-month follow-up and 12-month follow-up
  All participants were tested for microbial metabolites of vaginal secretions at 6-month follow-up and 12-month follow-up by LC-MS. Change in vaginal secretions metabolome from baseline to 12-month follow-up were assessed.
Serum metabolites testing at baseline | baseline
  All participants were tested for serum metabolites at enrollment by LC-MS. Measure abundances of serum metabolites, metabolic networks, and metabolic pathways activity.
Change in serum metabolome from baseline to 12-month follow-up assessments | 6-month follow-up and 12-month follow-up
  All participants were tested for microbial metabolites of serum at 6-month follow-up and 12-month follow-up by LC-MS. Change in serum metabolome from baseline to 12-month follow-up were assessed.

SECONDARY OUTCOMES:
vaginal cytokine testing at enrollment | Enrollment
  All participants were tested for IL-6 (pg/ml), IL-8 (pg/ml), IL-1β (pg/ml) and other cytokines in vaginal secretions at enrollment.
vaginal cytokine testing at 6-month follow-up | 6-month follow-up
  All participants were tested for IL-6 (pg/ml), IL-8 (pg/ml), IL-1β (pg/ml) and other cytokines in vaginal secretions at 6-month follow-up.
vaginal cytokine testing at 12-month follow-up | 12-month follow-up
  All participants were tested for IL-6 (pg/ml), IL-8 (pg/ml), IL-1β (pg/ml) and other cytokines in vaginal secretions at 12-month follow-up.
vaginal cytokine testing at 24-month follow-up | 24-month follow-up
  All participants were tested for IL-6 (pg/ml), IL-8 (pg/ml), IL-1β (pg/ml) and other cytokines in vaginal secretions at 24-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, PhD., Study Chair — Fujian Maternity and Child Health Hospital, Affiliated Hospital of Fujian Medical University
Locations (8):
- China (8):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Mindong Hospital of Ningde City, Ningde, Fujian
  - Quanzhou First Hospital Afflicated to Fujian Medical University, Quanzhou, Fujian
  - Xiamen Maternity and Child Health Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Zhangzhou affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Shunde Women's and Children's Hospital of Guangdong Medical University, Foshan, Guangdong
  - Maternal and Child Health Hospital of Shenzhen Province, Shenzhen, Guangdong
  - Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei